CLINICAL TRIAL: NCT06173284
Title: A Multi-Centered, Randomized, Double-Blinded, Placebo-Controlled Phase III Clinical Trial, to Evaluate the Efficacy and Safety of 611 (Recombinant Humanized Anti-interleukin-4 Receptor Alpha IgG4 Monoclonal Antibody) in Chinese Adults With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluation of 611(Recombinant Humanized Anti-interleukin-4 Receptor Alpha IgG4 Monoclonal Antibody) in Chinese Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-AD-III-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 611 (Experimental): Induction treatment period : subcutaneous injection, 611 600mg (loading dose, week 0) + 300mg Q2W (from Week 2 to Week 14, 7 cycles) Maintenance treatment period : subcutaneous injection, 611 300mg Q2W or Q4W
  Interventions: Drug: 611
- Placebo (Placebo Comparator): Induction treatment period : subcutaneous injection, placebo Q2W (from Week 0 to Week 14, 7 cycles) Maintenance treatment period : subcutaneous injection, 611 600mg (loading dose, week 16) + 300mg Q2W or Q4W
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: 611 — subcutaneous injection
  Arms: 611
Drug: Matching placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the efficacy of 611 in Chinese adults with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The maximum study duration was 64 weeks per participants, including a screening period of up to 4 weeks, a 52-week treatment period, and an 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and comply with the requirements of the study. and must participate voluntarily and sign the written informed consent.
2. Male or female adults ages 18 to 75 years old when signing the informed consent.
3. AD (according to Hanifin-Rajka Criteria) that had been present for at least 1 years before the screening visit.
4. Eczema Area and Severity Index (EASI) score greater than or equal to (>=) 16 at the screening and baseline visits.
5. Investigator's Global Assessment (IGA) score >=3 (on the 0 to 4 IGA scale, in which 3 was moderate and 4 was severe) at the screening and baseline visits.
6. Participants with >=10 percent (%) body surface area (BSA) of AD involvement at the screening and baseline visits.
7. Baseline Pruritus Numerical Rating Scale (NRS) average score for maximum itch intensity >=4.
8. Recent history (within 12 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments were otherwise medically inadvisable (e.g., because of important side effects or safety risks).
9. Have applied a stable dose of topical emollient (moisturizer) twice daily for at least the 7 consecutive days immediately before the baseline visit.
10. Female subjects of reproductive age (and their male partners) and male subjects (and their female partners) must use highly effective contraception throughout the study period and for at least 3 months after the last dose. The subjects had no plans to pregnancy, donate sperm or donate egg during the whole study period and for at least 3 months after the last dose.

Exclusion Criteria:

1. Presence of skin comorbidities that may interfere with study assessments
2. Presence of active endoparasitic infections; or suspected endoparasitic.
3. Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC).
4. History of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix at least 1 year, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin at least 1 year.
5. Active chronic or acute infection requiring treatment with systemic anti-infective therapy within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit.
6. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent infections, per investigator judgment.
7. Active TB, unless that was well documented that the participants had adequately treated.
8. Any medical condition that, in the opinion of the investigator, is serious or unstable and may affect the subject's safety and/or prevent the subject from completing the study
9. Treatment with topical drugs such as corticosteroids, topical calcineurin inhibitors, PDE inhibitors, or Janus kinase (JAK) inhibitors within 2 weeks before baseline;
10. The lab abnormalities at screening or baseline and not suitable for inclusion in the study judged by investigator;
11. Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
12. History of alcohol or drug abuse within 6 months before baseline.
13. History of hypersensitivity to 611 or their excipients.
14. Have been vaccinated with live (attenuated) vaccine within 2 months before baseline or planned during the study period;
15. Have used any investigational drug/treatment within 12 weeks before baseline;
16. Planned or anticipated major surgical procedure during the patient's participation in this study.
17. Pregnant or lactating women, or subjects with pregnancy or lactation plans during the study period.
18. Any reason which, in the opinion of investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Eczema Area and Severity Index (EASI) - 75 Response (>= 75% Improvement in Score From Baseline) at Week 16 | Baseline, Week 16
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants with Investigator's Global Assessment (IGA) Score of "0" or "1" and Improvement From Baseline of Greater Than or Equal to (>=) 2 Points From Baseline to Week 16 | Baseline，Week 16
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.

SECONDARY OUTCOMES:
Number of Participants With EASI-50 (>=50% Improvement From Baseline) | Baseline to Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants With EASI-90 (>=90% Improvement From Baseline) | Baseline to Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants Who Achieved >=4 Points/ >=3 Points With Improvement From Baseline in Weekly Average of Pruritus Numerical Rating Scale (NRS) Score From Baseline | Baseline to Week 60
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Percentage Change From Baseline in EASI Score | Baseline to Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Change From Baseline in Percent Body Surface Area (BSA) of AD Involvement | Baseline to Week 60
  BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and reported as a percentage of all major body sections combined. The reported percentage of BSA was combined percentage of all major body sections，with the higher scores reflecting the worse severity of AD.
Change From Baseline in Weekly Average of Pruritus NRS | Baseline to Week 60
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score | Baseline to Week 60
  The DLQI was a validated questionnaire used to measure the impact of AD disease symptoms and treatment on health-related quality of life (QOL). DLQI consisting of a set of 10 questions which assess QOL over the past week. Responses to each questions were assessed on a scale of 0 to 3, where 0 is "not at all" and 3 is "very much". Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Change From Baseline in Patient Oriented Eczema Measure (POEM) | Baseline to Week 60
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a scale ranging from 0 to 4 (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, 4 = all days). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicated more severe disease and poor quality of life.
Percentage of patients having achieved EASI-75 at Week 16 who continue to exhibit EASI-75 at Week 52 (EASI-75 calculated relative to baseline EASI score) | Baseline to Week 52
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Percentage of patients having achieved IGA 0 or 1 and a ≥2-point improvement from Baseline at Week 16 who continue to exhibit an IGA 0 or 1 and a ≥2-point improvement from Baseline at Week 52 | Baseline to Week 52
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit. | Up to 60 Weeks
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.
Minimum concentration (Cmin) | Baseline to Week 60
  Minimum concentration (Cmin) of 611
Percentage of Participants With Anti-drug Antibodies and Neutralizing Antibodies. | Baseline to Week 60.
  Immunogenicity assessment will be based on Anti-drug Antibodies (ADAs) response and development of Neutralizing Antibodies (NABs). Percentage is calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-drug antibodies / number of evaluable participants * 100%.
Change in serum concentrations of Pharmacodynamics indicators. | Baseline to Week 60.
  Pharmacodynamics indicators.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No